CLINICAL TRIAL: NCT03862430
Title: A Phase II Double-blind, RandomizEd, Prospective, Placebo Controlled STudy of NanO2TM Combined With Radiation and Temozolomide in Patients With Newly-diagnosed Glioblastoma multiformE: RESTORE
Brief Title: A Study of NanO2™ Combined With Radiation and Temozolomide in Patients With Newly Diagnosed GBM
Acronym: RESTORE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NuvOx LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RESTORE-P2
Record Dates: First submitted 2019-03-01; First posted 2019-03-05 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-06

CONDITIONS: Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- NanO2TM (Experimental): NanO2TM infusion in conjunction with Radiation Treatment and temozolomide
  Interventions: Drug: NanO2TM
- Placebo (Placebo Comparator): Placebo Saline infusion in conjunction with Radiation Treatment and temozolomide
  Interventions: Drug: Placebo Saline Infusion

INTERVENTIONS:
Drug: NanO2TM — 0.1 mL/kg NanO2 infusion
  Other Names: Dodecafluoropentane emulsion (DDFPe)
  Arms: NanO2TM
Drug: Placebo Saline Infusion — Saline Infusion
  Other Names: 0.9N NaCl
  Arms: Placebo

SUMMARY:
This clinical trial is testing the safety and efficacy of NanO2TM administered via intravenous infusion in combination with standard radiation and chemotherapy.

NanO2TM is being developed to increase the amount of oxygen delivered to tumors which is hoped to increase the effectiveness of radiation therapy.

DETAILED DESCRIPTION:
All study participants will receive standard care for GBM including Temozolomide and radiation therapy. Subjects will be randomized on a 2 to 1 basis to receive either NanO2 infusions or saline infusions immediately prior to standard radiation therapy. Radiation therapy is performed 5 days a week for 6 weeks.

Radiation therapy is followed 28 days of recovery, and then six cycles of maintenance Temozolomide therapy on days 1 to 5 of six 28 day cycles.

Follow up will be every 3 months for 3 years, and then every 6 months for another 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed, newly diagnosed primary or secondary glioblastoma multiforme.
2. Treatment plan includes 60 Gy of focal radiation administered in 30 fractions, concurrently with temozolomide chemotherapy.
3. Manageable risks associated with potential radiation necrosis in the radiation field, based on size of the field and proximity to eloquent brain regions (as assessed by the investigator).
4. Aged 18 years and older.
5. Karnofsky Performance Status ≥ 70
6. Life expectancy of at least 3 months.
7. Able to undergo gadolinium-enhanced MRI (Gd-MRI) scans.
8. Baseline MRI performed within 7 days before starting study treatment while on a stable or decreasing glucocorticoid dose for at least 7 days before and during the imaging study.
9. Adequate hematologic, renal and hepatic function, as defined by:

   1. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
   2. Platelet count ≥ 75 x 109/L
   3. Hemoglobin ≥ 10.0 g/dl
   4. Serum creatinine < 1.5 x ULN
   5. Total bilirubin within normal limits (≤ 2.5 x ULN if Gilbert's syndrome)
   6. Aspartate transaminase (AST) and Alanine transaminase (ALT) < 2.5 x ULN
10. Women of childbearing potential or men with child-bearing potential partners (unless vasectomized) must agree to use a highly-effective method of birth control from study entry until 4 months after completing study therapy.
11. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria

1. Recurrent Glioblastoma
2. Prior treatment for glioblastoma apart from surgical resection.
3. Presence of multi-focal glioblastoma disease that cannot be encompassed into a radiation treatment field that would be safely treated to the prescribed radiation dose.
4. Presence of leptomeningeal disease that cannot be encompassed within a feasible and safe radiation field.
5. Intracranial bleeding, except for stable grade 1 hemorrhage or a post-operative bleed that is clearing.
6. Has not recovered from the adverse effects of surgical resection or biopsy, except for neurological deficits.
7. Subjects who have received any other investigational agent within 4 weeks before enrollment
8. Stroke or transient ischemic attack requiring hospitalization within 6 months before enrollment.
9. Myocardial infarction (MI) within 6 months before enrolment, unstable angina, New York Heart Association (NYHA) class II or greater congestive heart failure, or uncontrolled hypertension (systolic BP > 160 mmHg and/or diastolic BP > 100 mmHg).
10. Known History of Congenital long QT syndrome (12-lead EKG is not required).
11. Clinically significant chronic obstructive pulmonary disease or asthma.
12. Active major infection requiring treatment.
13. A history of other malignancies, except adequately treated non-melanoma skin cancer, curatively treated in-situ cancers or other solid tumors curatively treated with no evidence of disease for ≥ 2 years.
14. Known infection with human immunodeficiency virus or hepatitis B or C virus (testing is not required).
15. Current anticoagulant or antiplatelet therapy, except for prophylactic doses of low molecular weight heparins, low-dose aspirin, rivaroxaban (Xarelto®), apixaban (Eliquis®), or dabigatran (Pradaxa®).
16. History of allergic reactions attributed to compounds of similar chemical composition to NanO2.
17. Women who are pregnant or breast feeding.
18. Inability to comply with study procedures.
19. History or evidence of any other clinically significant condition that, in the opinion of the investigator, would pose a risk to subject safety or interfere with study procedures, evaluation or completion.
20. Known hypersensitivity to any temozolomide component or to dacarbazine (DTIC).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Estimated)
Dates: Start 2023-03-31 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | 22 months
  To determine progression free survival (PFS) in newly-diagnosed glioblastoma patients after treatment with NVX-108 in combination with radiation and temozolomide (TMZ)

SECONDARY OUTCOMES:
Overall Survival | 22 Months
  To determine overall survival (OS) in newly-diagnosed glioblastoma patients after treatment with NanO2TM at the RD in combination with radiation and temozolomide.Neuro-oncology (RANO) criteria
Response assessment by mRANO | 22 Months
  To determine the objective response rate to study therapy using the modified Response Assessment in Neuro-oncology (mRANO) criteria
Response assessment for pseudoprogression | 22 Months
  To determine the effect of NanO2 on the timing of pseudoprogression occurrence
To confirm that NanO2 re-oxygenation | 22 Months
  Via TOLD MRI, we measure the oxygenation level in tumor tissue, to confirmd NanO2 treatment causes the re-oxygenation of hypoxic tissue
To estimate the effect on the duration of functional independence | 22 Months
  To estimate the effect on the duration of functional independence, as measured by the periodic measurement of Karnofsky Performance Scale
Patient quality of life | 22 Months
  To measure NanO2 treatment's impact on patient quality of life (score) by using FACT-Br
Caregiver quality of life | 22 Months
  To measure NanO2 treatment's impact on caregiver quality of life (score) by using questionnaires form CQOLC

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Center for Neurosciences, Tucson, Arizona
  - University of Arizona, Tucson, Arizona
  - UC Irvine Health- Chao Family Comprehensive Cancer Center, Orange, California
  - Providence St. John's Cancer Institute, Santa Monica, California
  - Yale Cancer Center, New Haven, Connecticut
  - St. Francis Medical Center, OSF Healthcare, Peoria, Illinois
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Saint Luke's Cancer Institute, Kansas City, Missouri
  - Atlantic Health System, Summit, New Jersey
  - Duke University Medical Center, Durham, North Carolina
  - University Hospitals Seidman Cancer Center, Cleveland, Ohio
  - Inova Schar Cancer Institute, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: Undecided